CLINICAL TRIAL: NCT02317731
Title: Effect of Use of Straw on Tolerability and Quality of Split Dose 4l-PEG Preparation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1410014830
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Colon Cancer
Keywords: bowel preparation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine (No Intervention): Subjects will ingest the bowel preparation from a cup
- Straw (Experimental): Subjects will ingest the bowel preparation with a straw
  Interventions: Other: Straw

INTERVENTIONS:
Other: Straw — Bowel preparation ingestion with a straw
  Arms: Straw

SUMMARY:
The purpose of this study is to determine whether patients drinking their bowel preparation solution with a straw will have improved tolerability for ingestion of their bowel preparation solution and achieve a higher bowel preparation quality score than patients drinking their bowel preparation solution without a straw.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 y/o scheduled for elective outpatient colonoscopy

Exclusion Criteria:

* History of colonic surgery, Contra-indication for preparation (PEG solution), History of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Bowel preparation quality | 1 day
  Bowel preparation quality will be measured using a validated scoring system (Boston Bowel Preparation Score) for bowel preparation

SECONDARY OUTCOMES:
Tolerability will be measured by subjective survey including a 5-point scale and a visual analog scale filled by the subjects the day of the colonoscopy | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Louis A Chaptini, MD, Principal Investigator — Yale University
Locations (1):
- Section of Digestive Diseases, Temple Medical Center, New Haven, Connecticut, United States